CLINICAL TRIAL: NCT00607373
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Mipomersen as Add-on Therapy in Homozygous Familial Hypercholesterolemia Subjects
Brief Title: Study to Assess the Safety and Efficacy of ISIS 301012 (Mipomersen) in Homozygous Familial Hypercholesterolemia
Acronym: RADICHOL 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 301012CS5; 2005-003449-15 (EudraCT Number)
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Lipid Metabolism, Inborn Errors; Hypercholesterolemia, Autosomal Dominant; Hyperlipidemias; Metabolic Diseases; Hyperlipoproteinemia Type II; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Metabolic Disorder; Congenital Abnormalities; Hypercholesterolemia; Hyperlipoproteinemias; Dyslipidemias; Lipid Metabolism Disorders
Keywords: Apolipoprotein B; Homozygous Familial Hypercholesterolemia; LDL-receptor gene
MeSH Terms: conditions — Lipid Metabolism, Inborn Errors; Hyperlipoproteinemia Type II; Hyperlipidemias; Metabolic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Congenital Abnormalities; Hypercholesterolemia; Hyperlipoproteinemias; Dyslipidemias; Lipid Metabolism Disorders; Homozygous Familial Hypercholesterolemia | interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mipomersen (Experimental): Participants received mipomersen 200 mg as a subcutaneous injection once a week for 26 weeks.
  Interventions: Drug: mipomersen
- Placebo (Placebo Comparator): Participants received placebo as a subcutaneous injection once a week for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mipomersen — 200 mg mipomersen administered once a week for 26 weeks as a 1 mL subcutaneous injection. Subjects weighing less than 50 kg received a lower dose of 160 mg (0.8mL) mipomersen.
  Other Names: ISIS 301012; mipomersen sodium; Kynamro™
  Arms: Mipomersen
Drug: Placebo — 1 mL subcutaneous injection once a week for 26 weeks. Subjects weighing less than 50 kg received 0.8 mL subcutaneous injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mipomersen (ISIS 301012) in subjects with homozygous familial hypercholesterolemia on lipid-lowering therapy.

This study consisted of a 26-week treatment period and a 24-week post-treatment follow-up period. Following treatment and Week 28 evaluations, participants could elect to enroll in an open-label extension study (301012-CS6; NCT00694109). Participants who were not eligible or elected not to enroll in the open-label extension study or who discontinued during the 28-week treatment period were followed in this study for 24 weeks from administration of the last dose of study drug.

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is an autosomal dominant genetic disorder of lipoprotein metabolism characterized by markedly elevated low density lipoprotein (LDL), premature onset of atherosclerosis and development of xanthomata. Patients with homozygous familial hypercholesterolemia (HoFH) have a severe disease that presents in childhood with total cholesterol typically in the 650 to 1000 mg/dL range.

This was a randomized, double-blind, placebo-controlled study, which consisted of a 4-week screening period, 26 weeks of treatment, and a 24-week post- treatment follow-up period (with the exception of patients who enrolled in the open-label extension study, Study 301012-CS6; NCT00694109). Eligible patients were randomized in a 2:1 ratio to receive 200 mg mipomersen or matching volume placebo subcutaneous (SC) injections weekly. Patients who weighed <50 kg received a lower dose of 160 mg mipomersen or matching volume of placebo SC injections weekly. Patients were to have been on a stable (>=12 weeks) regimen of allowed lipid-lowering therapies at screening, and were required to remain on the same dose and regimen throughout the study.

Patients returned to the study center for clinical evaluation every other week during the first 4 weeks of treatment, once every 4 to 5 weeks for the remainder of the treatment period, and monthly during the post-treatment evaluation (follow-up) period. The primary endpoint assessment was at Week 28. Following treatment and Week 28 evaluations, eligible patients who tolerated the study drug could elect to enroll in the open-label extension study (Study 301012-CS6; NCT00694109). Patients who did not participate in the open-label extension study were required to return to the study center for clinical evaluation at least twice during the post-treatment follow-up period, including an end-of-study termination visit at the end of this 24-week period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Homozygous Familial Hypercholesterolemia (HoFH)
* Stable lipid-lowering therapy for 12 weeks
* Stable weight for 6 weeks
* Stable low fat diet for 8 weeks

Exclusion Criteria:

* Significant health problems in the recent past including heart attack, stroke, blood disorders, cancer, or digestive problems

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (10):
- United States (2):
  - Charlotte, North Carolina
  - Cincinnati, Ohio
- São Paulo, São Paulo, Brazil
- Canada (2):
  - Chicoutimi, Quebec
  - Ste Foy, Quebec
- Mistri Wing, Singapore
- South Africa (2):
  - Observatory
  - Parktown
- Taipei, Taiwan
- London, United Kingdom

REFERENCES:
- [Derived] Duell PB, Santos RD, Kirwan BA, Witztum JL, Tsimikas S, Kastelein JJP. Long-term mipomersen treatment is associated with a reduction in cardiovascular events in patients with familial hypercholesterolemia. J Clin Lipidol. 2016 Jul-Aug;10(4):1011-1021. doi: 10.1016/j.jacl.2016.04.013. Epub 2016 May 9. PMID 27578134
- [Derived] Santos RD, Raal FJ, Catapano AL, Witztum JL, Steinhagen-Thiessen E, Tsimikas S. Mipomersen, an antisense oligonucleotide to apolipoprotein B-100, reduces lipoprotein(a) in various populations with hypercholesterolemia: results of 4 phase III trials. Arterioscler Thromb Vasc Biol. 2015 Mar;35(3):689-99. doi: 10.1161/ATVBAHA.114.304549. Epub 2015 Jan 22. PMID 25614280
- [Derived] Raal FJ, Santos RD, Blom DJ, Marais AD, Charng MJ, Cromwell WC, Lachmann RH, Gaudet D, Tan JL, Chasan-Taber S, Tribble DL, Flaim JD, Crooke ST. Mipomersen, an apolipoprotein B synthesis inhibitor, for lowering of LDL cholesterol concentrations in patients with homozygous familial hypercholesterolaemia: a randomised, double-blind, placebo-controlled trial. Lancet. 2010 Mar 20;375(9719):998-1006. doi: 10.1016/S0140-6736(10)60284-X. PMID 20227758

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-one patients were screened and fifty-one randomized. Eligible patients were randomized in a 2:1 ratio to receive 200 mg mipomersen or matching volume placebo subcutaneous (SC) injections weekly.
Period: Treatment Period
Arm/Group | Placebo | Mipomersen
Started | 17 | 34
Completed | 17 (16 enrolled in open-label extension study NCT00694109) | 28 (23 enrolled in open-label extension study NCT00694109)
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Follow-up Period
Arm/Group | Placebo | Mipomersen
Started | 1 (Participants enrolled in the open-label extension (NCT00694109) or continued in the follow-up period) | 11 (Participants enrolled in the open-label extension (NCT00694109) or continued in the follow-up period)
Completed | 0 | 6
Not Completed | 1 | 5
Not completed — Other | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mipomersen | Total
Number analyzed (Participants) | 17 | 34 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (14.1) | 30.4 (11.5) | 31.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 19 | 29
  Male | 7 | 15 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 16 | 29 | 45
Race/Ethnicity, Customized [Number; unit: participants]
  White | 13 | 25 | 38
  Asian | 3 | 8 | 11
  Black | 1 | 1 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.32 (4.41) | 25.97 (5.81) | 26.08 (5.34)
Waist/hip ratio [Mean (Standard Deviation); unit: ratio] | 0.83 (0.07) | 0.85 (0.06) | 0.84 (0.07)
Metabolic syndrome [Number; unit: participants] — Yes if 3 or more risk factors are present:
  1) Abdominal obesity 2) Triglycerides >=150 mg/dl * 3) High density lipoprotein cholesterol (men <40 mg/dl) (women <50 mg/dl) * 4) Systolic blood pressure >=130 or diastolic >=85 mmHg * 5) Fasting glucose >=100 mg/dl *
  * = or on medication for condition
  participants
    No | 16 | 27 | 43
    Yes | 1 | 7 | 8
Tobacco Use [Number; unit: participants]
  Current | 3 | 7 | 10
  Non-current | 3 | 4 | 7
  Never | 11 | 23 | 34
Alcohol Use [Number; unit: participants]
  Current | 6 | 14 | 20
  Non-current | 3 | 3 | 6
  Never | 8 | 17 | 25
Fasting serum insulin [Mean (Standard Deviation); unit: microIU/mL] | 9.72 (5.98) | 11.54 (14.78) | 10.93 (12.51)
Fasting hemoglobin A1c [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 5.47 (0.22) | 5.34 (0.37) | 5.38 (0.33)
Weight [Number; unit: participants] — Participants who weighed <50 kg received the lower dose of 160 mg mipomersen or matching placebo. All other patients received a dose of 200 mg or matching placebo.
  participants
    <50 kg | 2 | 4 | 6
    >=50 kg | 15 | 30 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Primary Efficacy Time Point
Description: LDL-C was measured in mg/dL. Samples were taken following an overnight fast. For patients with triglycerides <400 mg/dL, LDL-C was obtained using Friedewald's calculation; and for patients with triglycerides >=400 mg/dL, LDL-C was directly measured by the central laboratory using ultracentrifugation. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. If the Study Day 1 and screening LDL-C values were >12% different (relative to the maximum value), then the screening value was not used, because the Study Day 1 value represents the best estimate of the patient's condition at the beginning of study drug administration. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: Baseline (the average of the screening and Day 1 pre-treatment assessments) and the Primary Efficacy Time point (PET) up to week 28
Population: Full analysis set (FAS). The FAS, which represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9, consists of treated participants with a valid baseline and at least one post-baseline LDL-C measure.
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
percentage of baseline | -3.31 (17.06) | -24.66 (19.85)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Based upon prior clinical study experience with mipomersen, it was estimated that the standard deviation of the percent change in LDL-C is approximately 22%. With 15 patients in the control group and 30 patients in the mipomersen-treated group, this study would have at least 80% power to detect a 20 percentage point difference between the 2 treatment groups. Fifty-one patients were enrolled to allow for patient withdrawals and potential exclusions from analysis sets; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Statistical significance was concluded if p≤0.05

2. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo-B) at Primary Efficacy Time Point
Description: Apo-B was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
percentage of baseline | -2.54 (12.56) | -26.77 (17.04)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Inflation of type 1 error was controlled by specifying a small number of secondary parameters and a sequential inferential approach in which inferential conclusions about each successive parameter required statistical significance of the prior one

3. Secondary Outcome: Apo-B at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: Baseline (the average of the screening and Day 1 pre-treatment assessments) and the Primary Efficacy Time point (PET) up to week 28 )
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
mg/dL
  Baseline | 259.2 (84.4) | 283.1 (78.4)
  PET | 252.6 (85.0) | 205.4 (70.0)

4. Secondary Outcome: Percentage Change From Baseline in Total Cholesterol at Primary Efficacy Time Point (PET)
Description: Total cholesterol was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
percentage of baseline | -1.98 (14.82) | -21.20 (17.69)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Inferential conclusions about this parameter require statistical significance of the previous secondary outcome measure (i.e., percent change from baseline in Apo B at PET)

5. Secondary Outcome: Total Cholesterol at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
mg/dL
  Baseline | 460.5 (132.0) | 502.4 (144.5)
  PET | 452.1 (144.6) | 389.7 (125.3)

6. Primary Outcome: LDL-C at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
mg/dL
  Baseline | 400.2 (141.5) | 438.9 (138.6)
  PET | 388.2 (150.5) | 326.2 (121.3)

7. Secondary Outcome: Percentage Change From Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at Primary Efficacy Time Point (PET)
Description: Non-HDL-C was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
percentage of baseline | -2.90 (16.32) | -24.50 (19.17)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Inferential conclusions about this parameter require statistical significance of the previous secondary outcome measure (i.e., percent change from baseline in total cholesterol at PET)

8. Secondary Outcome: Non-HDL-C at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
mg/dL
  Baseline | 418.9 (144.5) | 464.3 (145.4)
  PET | 409.1 (156.6) | 345.8 (126.6)

9. Other Pre Specified Outcome: Percentage Change From Baseline in Triglycerides at Primary Efficacy Time Point (PET)
Description: Triglycerides were measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
percentage of baseline | 0.9 [-25.0 to 29.5] | -17.5 [-36.0 to -4.8]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.013, Wilcoxon rank sum test — Statistical significance was concluded if p ≤0.05

10. Other Pre Specified Outcome: Triglycerides at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
mg/dL
  Baseline | 92 [80 to 105] | 91 [73 to 141]
  PET | 85 [65 to 117] | 76 [52 to 116]

11. Other Pre Specified Outcome: Percentage Change From Baseline in Lipoprotein(a) at Primary Efficacy Time Point (PET)
Description: Lipoprotein(a) was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
percentage of baseline | -7.87 (21.87) | -31.10 (23.02)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — Statistical significance was concluded if p ≤0.05

12. Other Pre Specified Outcome: Lipoprotein(a) at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
mg/dL
  Baseline | 66.3 (53.1) | 64.3 (41.0)
  PET | 61.6 (52.6) | 43.8 (32.1)

13. Other Pre Specified Outcome: Percentage Change From Baseline in Very-Low-Density Lipoprotein Cholesterol (VLDL-C) at Primary Efficacy Time Point (PET)
Description: VLDL-C was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
percentage of baseline | 2.3 [-25.0 to 28.6] | -17.3 [-37.1 to -3.0]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.009, Wilcoxon rank sum test — Statistical significance was concluded if p ≤0.05

14. Other Pre Specified Outcome: VLDL-C at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
mg/dL
  Baseline | 18 [16 to 21] | 18 [15 to 28]
  PET | 17 [13 to 23] | 15 [10 to 23]

15. Other Pre Specified Outcome: Change From Baseline in Ratio of Low-density Lipoprotein Cholesterol (LDL-C) to High-density Lipoprotein Cholesterol (HDL-C) at Primary Efficacy Time Point (PET)
Description: LDL-C and HDL-C were measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
percentage of baseline | -6.22 (18.81) | -34.32 (21.00)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Statistical significance was concluded if p ≤0.05

16. Other Pre Specified Outcome: Ratio of LDL-C to HDL-C at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
ratio
  Baseline | 12.14 (7.675) | 13.02 (6.115)
  PET | 11.37 (7.095) | 8.13 (3.921)

17. Other Pre Specified Outcome: Percent Change From Baseline in Apolipoprotein A1 (Apo-A1) at Primary Efficacy Time Point (PET)
Description: Apo-A1 was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
percentage of baseline | 5.35 (10.63) | 9.27 (17.59)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.328, t-test, 2 sided — Statistical significance was concluded if p ≤0.05

18. Other Pre Specified Outcome: Apo-A1 at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
mg/dL
  Baseline | 118.6 (33.0) | 111.5 (27.9)
  PET | 124.5 (34.9) | 118.8 (20.5)

19. Other Pre Specified Outcome: Percentage Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at Primary Efficacy Time Point (PET)
Description: HDL-C was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
percentage of baseline | 4.1 [-2.0 to 13.2] | 14.8 [3.3 to 27.0]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.035, Wilcoxon rank sum test — Statistical significance was concluded if p ≤0.05

20. Other Pre Specified Outcome: HDL-C at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 17 | 34
mg/dL
  Baseline | 38 [27 to 49] | 35 [32 to 44]
  PET | 43 [28 to 53] | 43 [37 to 48]

ADVERSE EVENTS:
Time Frame: Day 1 to week 28. On-treatment AEs started on/after the first study drug dose and on/before the end of the treatment period. The treatment period was the time study drug was administered until the later of the PET or 14 days after last study drug dose.
Description: The Safety Set includes all randomized patients who receive at least 1 injection of the study treatment. In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Placebo | Mipomersen
Serious Adverse Events (participants affected / at risk) | 1/17 | 2/34
Other Adverse Events (participants affected / at risk) | 13/17 | 30/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | Mipomersen (N=34)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | Mipomersen (N=34)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1
Cardiac discomfort (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 6
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 4
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 3
Injection site anaesthesia (General disorders) | 0 | 1
Injection site discolouration (General disorders) | 0 | 10
Injection site discomfort (General disorders) | 0 | 3
Injection site erythema (General disorders) | 1 | 19
Injection site haematoma (General disorders) | 2 | 12
Injection site haemorrhage (General disorders) | 0 | 1
Injection site induration (General disorders) | 0 | 2
Injection site inflammation (General disorders) | 0 | 1
Injection site irritation (General disorders) | 1 | 1
Injection site macule (General disorders) | 0 | 5
Injection site oedema (General disorders) | 0 | 2
Injection site pain (General disorders) | 1 | 12
Injection site pallor (General disorders) | 0 | 2
Injection site papule (General disorders) | 0 | 4
Injection site paraesthesia (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 1 | 10
Injection site rash (General disorders) | 0 | 2
Injection site recall reaction (General disorders) | 0 | 1
Injection site swelling (General disorders) | 0 | 4
Injection site warmth (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Red blood cell macrocytes present (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Facial palsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 5
Neuralgia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Galactorrhoea (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication for a multi-centre trial must address all centers. Institution will submit for review a proposed publication or presentation at least 60 days prior to submission date. Sponsor has the right to delay publication or presentation for not more than 6 months (contracts have variable timeframes) to address patent applications. Sponsor also has the right to demand in writing the deletion of confidential information, as long as such removal will not preclude publication.